CLINICAL TRIAL: NCT00045786
Title: A Multi-center, An Open Label, Dose-Escalation Study to Determine the Safety and Preliminary Efficacy of CC-1088 in the Treatment for Myelodysplastic Syndromes
Brief Title: Study to Determine the Safety and Preliminary Efficacy of CC-1088 in the Treatment of Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-1088-MDS-801-001
Record Dates: First submitted 2002-09-09; First posted 2002-09-11 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

ARMS (4):
- 400 mg CC-1088 (Experimental)
  Interventions: Drug: CC-1088
- 800 mg CC-1088 (Experimental)
  Interventions: Drug: CC-1088
- 1200 mg CC-1088 (Experimental)
  Interventions: Drug: CC-1088
- 1500 mg CC-1088 (Experimental)
  Interventions: Drug: CC-1088

INTERVENTIONS:
Drug: CC-1088 — 400 mg/day (200 mg orally twice a day) 800 mg/day (400 mg orally twice a day) 1200 mg/day (600 mg orally twice a day) 1500 mg/day (500 mg orally three times daily)

SUMMARY:
The primary objective of the study is to assess the safety of CC-1088 to patients with myelodysplastic syndromes (MDS).

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must have a diagnosis of MDS of at least 12 weeks that is not therapy related.
* Age ≥ 18 at the time of signing informed consent
* Patient must be able to adhere to the study visit schedule and other protocol requirements.
* Patient must understand and voluntarily sign an informed consent document.
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test.
* Sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).
* Women must not be pregnant or lactating.

Exclusion Criteria

* Pregnant and lactating women and WCBP who are not using adequate contraception.
* Myelosclerosis (or myelofibrosis) occupying >30% of marrow space
* Patients with iron deficiency (e.g., absent bone marrow iron store). If a marrow aspirate is not evaluable for storage iron, transferrin saturation must be 220% and serum femtin not less than 50 ng/mL.
* Patients with uncorrected Bl2 or folate deficiency.
* Patients with contributing causes of anemia such as autoimmune or heredity, hemolytic disorders, or GI blood loss.
* Patients with a history of malignancy, except basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ.
* Patients with clinically significant, symptomatic and unstable pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal or genitourinary system diseases unrelated to their underlying hematologic disorder.
* Life-threatening or active infection requiring parenteral antibiotic therapy or other serious concurrent illness.
* Patients who have a history of testing positive for Hepatitis B surface antigenemia,'Hepatitis C, or HIV.
* Inadequate organ hction: renal insufficiency [serum creatinine levels >1.5 x upper limit of normal (ULN)] or hepatic impairment (bilirubin 22 mg/dL or AST/ALT 22 x ULN).
* Patients may not have received another investigational study drug within 30 days of entry in the present study.
* Requirement for ongoing therapy with corticosteroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2001-10; Primary Completion 2001-12 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, Study Director — Celgene Corporation
Locations (1):
- Rush-Presbyterian-St Luke's Medical Center, Chicago, Illinois, United States